CLINICAL TRIAL: NCT03021187
Title: Efficacy and Safety of Oral Semaglutide Versus Placebo in Subjects With Type 2 Diabetes Mellitus Treated With Insulin. A 52-week, Randomised, Double-blind, Placebo-controlled Trial (PIONEER 8 - Insulin add-on)
Brief Title: Efficacy and Safety of Oral Semaglutide Versus Placebo in Subjects With Type 2 Diabetes Mellitus Treated With Insulin
Acronym: PIONEER 8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4280; 2016-000988-16 (EudraCT Number); U1111-1180-3637 (Other: World Health Organization (WHO)); JapicCTI-173508 (Other: JAPIC)
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Semaglutide 3 mg (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 3 mg + 7 mg (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 3 mg + 7 mg + 14 mg (Experimental)
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Oral semaglutide administered once-daily for 52 weeks as an add-on to the subjects' pre-trial insulin treatment
  Arms: Semaglutide 3 mg
Drug: semaglutide — Oral semaglutide (3 mg followed by 7 mg) administered once-daily for 52 weeks as an add-on to the subjects' pre-trial insulin treatment
  Arms: Semaglutide 3 mg + 7 mg
Drug: semaglutide — Oral semaglutide (3 mg followed by 7 mg and finally 14 mg) administered once-daily for 52 weeks as an add-on to the subjects' pre-trial insulin treatment
  Arms: Semaglutide 3 mg + 7 mg + 14 mg
Drug: placebo — Oral semaglutide placebo administered once-daily for 52 weeks as an add-on to the subjects' pre-trial insulin treatment
  Arms: Placebo

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate the efficacy and safety of oral semaglutide versus placebo in subjects with Type 2 Diabetes Mellitus treated with insulin. All subjects should continue their pre-trial insulin therapy (basal, basal-bolus or premixed regimen including combinations of soluble insulins) throughout the trial. Subjects treated with metformin in addition to insulin treatment must continue their metformin treatment throughout the entire trial.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial. - Male or female, age above or equal to 18 years at the time of signing informed consent. For Japan only: Male or female, age above or equal to 20 years at the time of signing informed consent. - Diagnosed with type 2 diabetes mellitus 90 days or more prior to the day of screening. - HbA1c (glycosylated haemoglobin) of 7.0-9.5% (53-80 mmol/mol) (both inclusive). - Stable treatment with one of the following insulin regimens (minimum 10 IU/day) 90 or more days prior to the day of screening. Maximum 20% change in total daily dose is acceptable: (1) Basal insulin alone or (2) Basal and bolus insulin in any combination or (3) Premixed insulin including combinations of soluble insulins Exclusion Criteria: - Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice). For Greece only: adequate contraceptive measures are defined as combined hormonal contraception (containing oestrogen and progesterone), which suppress ovulation (oral, intravaginal, percutaneous), progesterone-only hormonal contraception which suppress ovulation (oral, injectable, implantable), intrauterine device, hormone-releasing intrauterine system, bilateral tubal occlusion, partner with vasectomy, sexual abstinence. For Japan only: Adequate contraceptive measures are abstinence (not having sex), diaphragm, condom (by the partner), intrauterine device, sponge, spermicide or oral contraceptives. For Canada only: adequate contraceptive measures are defined as combined hormonal contraception (containing oestrogen and progesterone), which suppress ovulation (oral, intravaginal, percutaneous), progesterone-only hormonal contraception which suppress ovulation (oral, injectable, implantable), intrauterine device, hormone-releasing intrauterine system, bilateral tubal occlusion, partner with vasectomy, sexual abstinence - Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol. - Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN 2) or Medullary Thyroid Carcinoma (MTC). - History of pancreatitis (acute or chronic). - History of major surgical procedures involving the stomach and potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery). - Any of the following: myocardial infarction (MI), stroke or hospitalisation for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation. - Classified as being in New York Heart Association (NYHA) Class IV. - Planned coronary, carotid or peripheral artery revascularisation known on the day of screening. - Renal impairment defined as estimated Glomerular Filtration Rate (eGFR) less than 60 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI). - Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening. An exception is short-term change of insulin treatment for acute illness for a total of 14 days or less. - Known hypoglycaemic unawareness according to Clarke's questionnaire. - Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to randomisation. - History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and carcinoma in situ). - Subjects with alanine aminotransferase (ALT) more than 2.5 x upper normal limit (UNL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (47):
  - Novo Nordisk Investigational Site, Anniston, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Fountain Hills, Arizona
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Riverside, California
  - Novo Nordisk Investigational Site, Van Nuys, California
  - Novo Nordisk Investigational Site, Vista, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Franklin, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Natchitoches, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Lansdale, Pennsylvania
  - Novo Nordisk Investigational Site, Summerville, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Mesquite, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Murray, Utah
  - Novo Nordisk Investigational Site, Winchester, Virginia
- Canada (7):
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Moncton, New Brunswick
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Waterloo, Ontario
- France (12):
  - Novo Nordisk Investigational Site, Besançon
  - Novo Nordisk Investigational Site, Bourgoin
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, La Roche-sur-Yon
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Coudray
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Vénissieux
- Greece (5):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Ioannina
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Piraeus
  - Novo Nordisk Investigational Site, Thessaloniki
- India (11):
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kozhikode, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Kolkata
- Japan (17):
  - Novo Nordisk Investigational Site, Amagasaki-shi, Hyogo
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi, Kanagawa
  - Novo Nordisk Investigational Site, Iruma-shi, Saitama
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kumamoto
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Saga-shi, Saga
  - Novo Nordisk Investigational Site, Sapporo
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Ube-shi, Yamaguchi
- Mexico (2):
  - Novo Nordisk Investigational Site, Durango
  - Novo Nordisk Investigational Site, San Luis Potosí City
- Poland (4):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Puławy
- Novo Nordisk Investigational Site, Manatí, Puerto Rico
- Russia (4):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Zinman B, Aroda VR, Buse JB, Cariou B, Harris SB, Hoff ST, Pedersen KB, Tarp-Johansen MJ, Araki E; PIONEER 8 Investigators. Efficacy, Safety, and Tolerability of Oral Semaglutide Versus Placebo Added to Insulin With or Without Metformin in Patients With Type 2 Diabetes: The PIONEER 8 Trial. Diabetes Care. 2019 Dec;42(12):2262-2271. doi: 10.2337/dc19-0898. Epub 2019 Sep 17. PMID 31530667
- [Derived] Pratley RE, Crowley MJ, Gislum M, Hertz CL, Jensen TB, Khunti K, Mosenzon O, Buse JB. Oral Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Glucose-Lowering Medication: PIONEER Subgroup Analyses. Diabetes Ther. 2021 Apr;12(4):1099-1116. doi: 10.1007/s13300-020-00994-9. Epub 2021 Mar 4. PMID 33660198
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 111 sites in 9 countries: Canada (7), France (10), Greece (6), India (9), Japan (18), Mexico (2), Poland (4), Russian Federation (5) and United States (48). Following sites were approved by the IRB/IEC but didn't randomise subjects: France (2), India (1), Japan (1) and United States (3).
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 3 mg: Participants were to take oral semaglutide 3 mg tablets once-daily from week 0 to week 52.
- Oral Semaglutide 7 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 52: 3 mg from week 0 to week 4 and 7 mg from week 4 to week 52.
- Oral Semaglutide 14 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 52: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 8 to week 52.
- Placebo: Participants were to take oral semaglutide placebo tablets once-daily for a period of 52 weeks.
Period: Overall Study
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Started | 184 | 182 | 181 | 184
Exposed | 184 | 181 | 181 | 184
Full Analysis Set (FAS) | 184 | 182 | 181 | 184
Safety Analysis Set (SAS) | 184 | 181 | 181 | 184
Completed | 174 | 173 | 175 | 175
Not Completed | 10 | 9 | 6 | 9
Not completed — Death | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 2 | 5
Not completed — Lost to Follow-up | 10 | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo | Total
Number analyzed (Participants) | 184 | 182 | 181 | 184 | 731
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9) | 60 (10) | 61 (10) | 60 (10) | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 79 | 96 | 79 | 336
  Male | 102 | 103 | 85 | 105 | 395
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was recorded as 'Not Applicable' for France as per local regulation.
  Participants
    White | 89 | 95 | 94 | 98 | 376
    Black or African American | 15 | 10 | 11 | 13 | 49
    Asian | 66 | 66 | 66 | 65 | 263
    American Indian or Alaska native | 1 | 0 | 1 | 0 | 2
    Native Hawaiian or other Pacific | 0 | 0 | 0 | 0 | 0
    Other | 1 | 1 | 1 | 0 | 3
    Not applicable | 12 | 10 | 8 | 8 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity was recorded as 'Not Applicable' for France as per local regulation.
  Participants
    Hispanic or Latino | 18 | 24 | 30 | 25 | 97
    Non hispanic or Latino | 154 | 148 | 143 | 150 | 595
    Not applicable | 12 | 10 | 8 | 9 | 39
HbA1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — Glycosylated haemoglobin
  Percentage of HbA1c | 8.2 (0.7) | 8.2 (0.7) | 8.2 (0.7) | 8.2 (0.7) | 8.2 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Week 26)
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at week 26. The endpoint was evaluated based on data from the in-trial observation period. In-trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any. The endpoint was also analysed based on data from the on-treatment without rescue medication observation period. On-treatment without rescue medication observation period started at the date of the first dose of trial product and includes the period after initiation of rescue medication, if any, and excludes the period after premature trial discontinuation, if any.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Percentage of HbA1c
  In-trial: number analyzed (Participants) | 176 | 174 | 173 | 176
  In-trial | -0.5 (1.0) | -1.0 (1.1) | -1.3 (1.1) | -0.1 (0.9)
  On-treatment without rescue medication: number analyzed (Participants) | 162 | 157 | 146 | 161
  On-treatment without rescue medication | -0.6 (1.1) | -1.1 (1.0) | -1.4 (0.9) | -0.1 (0.8)
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an analysis of covariance (ANCOVA) model with treatment, strata, interaction strata and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand); p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.5, 95% CI 2-sided [-0.7 to -0.3] — Oral semaglutide 3mg - Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment, strata, interaction strata and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.9, 95% CI 2-sided [-1.1 to -0.7] — Oral semaglutide 7 mg - Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.2, 95% CI 2-sided [-1.4 to -1.0] — Oral semaglutide 14 mg - Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 3 mg vs Placebo; The analysis was based on a mixed model for repeated measurements (MMRM) that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, region, strata and interaction strata as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the on-treatment without rescue medication observation period. The estimated treatment effect excludes the effect of any rescue medication and any effect after premature trial product discontinuation (hypothetical estimand); p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.6, 95% CI 2-sided [-0.7 to -0.4] — Oral semaglutide 3 mg - Placebo
Statistical Analysis 5: Comparison: Oral Semaglutide 7 mg vs Placebo; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, region, strata and the interaction strata as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.0, 95% CI 2-sided [-1.2 to -0.8] — Oral semaglutide 7 mg - Placebo
Statistical Analysis 6: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 1, analysis 5]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -1.4, 95% CI 2-sided [-1.6 to -1.2] — Oral semaglutide 14 mg - Placebo

2. Secondary Outcome: Change in Body Weight (Week 26)
Description: Change from baseline (week 0) in body weight was evaluated at week 26. The endpoint was evaluated based on data from the in-trial observation period. In-trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any. The endpoint was also evaluated based on data from the on-treatment without rescue medication observation period. It started at the date of first dose of trial product and excluded the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Kg
  In trial: number analyzed (Participants) | 177 | 174 | 173 | 177
  In trial | -1.4 (3.1) | -2.6 (5.2) | -3.7 (4.0) | -0.5 (2.5)
  On-treatment without rescue medication: number analyzed (Participants) | 163 | 157 | 146 | 162
  On-treatment without rescue medication | -1.5 (3.1) | -3.0 (3.7) | -3.9 (3.6) | -0.5 (2.4)
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment, strata, interaction strata and region as categorical fixed effects and baseline body weight value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0392, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.9, 95% CI 2-sided [-1.8 to -0.0] — Oral semaglutide 3 mg - Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -2.0, 95% CI 2-sided [-3.0 to -1.0] — Oral semaglutide 7 mg - Placebo
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -3.3, 95% CI 2-sided [-4.2 to -2.3] — Oral semaglutide 14 mg - Placebo
Statistical Analysis 4: Comparison: Oral Semaglutide 3 mg vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p = 0.0111, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -0.9, 95% CI 2-sided [-1.6 to -0.2] — Oral semaglutide 3 mg - Placebo
Statistical Analysis 5: Comparison: Oral Semaglutide 7 mg vs Placebo; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, region, strata and the interaction strata as categorical fixed effects and the baseline body weight value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -2.5, 95% CI 2-sided [-3.2 to -1.8] — Oral semaglutide 7 mg - Placebo
Statistical Analysis 6: Comparison: Placebo; [analysis description as in outcome 2, analysis 5]; Test type: Superiority — [test comment as in outcome 1, analysis 4]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0 (superiority); Mean treatment difference = -3.7, 95% CI 2-sided [-4.4 to -3.0] — Oral semaglutide 14 mg - Placebo

3. Secondary Outcome: Change in HbA1c (Week 52)
Description: Change from baseline (week 0) in HbA1c to week 52. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 173 | 169 | 168 | 172
Percentage of HbA1c | -0.6 (1.0) [lower limit 1.0] | -0.9 (1.1) [lower limit 1.1] | -1.2 (1.0) [lower limit 1.0] | -0.2 (0.8) [lower limit 0.8]

4. Secondary Outcome: Change in Body Weight (kg) (Week 52)
Description: Change from baseline (week 0) in body weight to week 52. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 174 | 171 | 170 | 173
Kg | -0.9 (3.9) [lower limit 3.9] | -2.2 (5.2) [lower limit 5.2] | -3.8 (5.8) [lower limit 5.8] | 0.5 (3.2) [lower limit 3.2]

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG to week 26 and week 52. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
mmol/L
  Week 26: number analyzed (Participants) | 175 | 173 | 173 | 175
  Week 26 | -0.45 (3.35) | -1.14 (3.08) | -1.36 (2.72) | 0.51 (2.84)
  Week 52: number analyzed (Participants) | 172 | 168 | 169 | 172
  Week 52 | -0.81 (3.21) | -1.12 (2.91) | -1.60 (2.65) | -0.09 (2.97)

6. Secondary Outcome: Change in Self-measured Plasma Glucose (SMPG) Mean 7-point Profile
Description: Change from baseline (week 0) in self-measured plasma glucose (SMPG) mean 7-point profile to week 26 and week 52. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. Mean 7-point profile was defined as the area under the profile, calculated using the trapezoidal method, divided by the measurement time. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
mmol/L
  Week 26: number analyzed (Participants) | 171 | 164 | 159 | 167
  Week 26 | -1.2 (2.3) | -1.8 (2.4) | -2.0 (2.2) | -0.3 (2.7)
  Week 52: number analyzed (Participants) | 163 | 157 | 157 | 159
  Week 52 | -1.6 (2.5) | -1.7 (2.4) | -2.0 (2.1) | -0.9 (2.4)

7. Secondary Outcome: Change in SMPG Mean Postprandial Increment Over All Meals
Description: Change from baseline (week 0) in SMPG mean postprandial increment over all meals to week 26 and week 52. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
mmol/L
  Week 26: number analyzed (Participants) | 170 | 161 | 158 | 167
  Week 26 | -0.3 (2.3) | -0.8 (2.6) | -1.2 (2.5) | -0.1 (2.8)
  Week 52: number analyzed (Participants) | 161 | 153 | 156 | 155
  Week 52 | -0.3 (2.3) | -0.7 (2.3) | -0.7 (2.3) | -0.3 (2.4)

8. Secondary Outcome: Change in Body Weight (Percentage)
Description: Relative change from baseline (week 0) in body weight (%) was evaluated at weeks 26 and 52.The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Percentage change
  Week 26: number analyzed (Participants) | 177 | 174 | 173 | 177
  Week 26 | -1.73 (3.34) | -3.11 (5.66) | -4.30 (4.57) | -0.47 (3.02)
  Week 52: number analyzed (Participants) | 174 | 171 | 170 | 173
  Week 52 | -1.18 (4.17) | -2.54 (5.77) | -4.42 (6.07) | 0.65 (3.72)

9. Secondary Outcome: Change in Body Mass Index
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at weeks 26 and 52. BMI was calculated based on body weight and height based on the formula: BMI kg/m^2 = body weight (kg)/(Height (m) x Height (m)). Data based on in-trial observation period is presented. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
kg/m^2
  Week 26: number analyzed (Participants) | 177 | 174 | 173 | 177
  Week 26 | -0.5 (1.1) | -1.0 (1.7) | -1.4 (1.5) | -0.2 (0.9)
  Week 52: number analyzed (Participants) | 174 | 171 | 170 | 173
  Week 52 | -0.3 (1.4) | -0.8 (1.8) | -1.4 (2.1) | 0.2 (1.2)

10. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at weeks 26 and 52.The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
cm
  Week 26: number analyzed (Participants) | 176 | 173 | 173 | 176
  Week 26 | -0.9 (4.1) | -2.3 (5.1) | -3.6 (4.9) | -0.6 (3.6)
  Week 52: number analyzed (Participants) | 172 | 171 | 170 | 173
  Week 52 | -0.8 (4.8) | -2.3 (5.1) | -4.0 (6.8) | 0.3 (4.1)

11. Secondary Outcome: Change in Total Cholesterol - Ratio to Baseline
Description: Change from baseline in total cholesterol (mmol/L) is presented as ratio to baseline at week 26 and week 52. Results are based on the data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Ratio of total cholesterol
  Week 26: number analyzed (Participants) | 176 | 172 | 170 | 175
  Week 26 | 0.99 (15.5) | 0.95 (18.7) | 0.95 (17.3) | 1.03 (15.4)
  Week 52: number analyzed (Participants) | 173 | 167 | 167 | 170
  Week 52 | 0.98 (18.2) | 0.97 (19.2) | 0.95 (18.1) | 1.00 (17.6)

12. Secondary Outcome: Change in LDL Cholesterol - Ratio to Baseline
Description: Change from baseline in LDL cholesterol (mmol/L) is presented as ratio to baseline at week 26 and week 52. Results are based on the data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Ratio of LDL cholesterol
  Week 26: number analyzed (Participants) | 176 | 172 | 170 | 175
  Week 26 | 0.98 (27.1) | 0.93 (30.2) | 0.93 (24.5) | 1.03 (25.9)
  Week 52: number analyzed (Participants) | 172 | 167 | 167 | 169
  Week 52 | 0.97 (29.2) | 0.96 (29.4) | 0.95 (27.6) | 1.00 (28.3)

13. Secondary Outcome: Change in HDL Cholesterol - Ratio to Baseline
Description: Change from baseline (week 0) in HDL cholesterol (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Ratio of HDL cholesterol
  Week 26: number analyzed (Participants) | 176 | 172 | 170 | 175
  Week 26 | 1.00 (13.5) | 0.98 (13.5) | 0.98 (16.7) | 1.01 (13.0)
  Week 52: number analyzed (Participants) | 172 | 167 | 167 | 170
  Week 52 | 1.01 (14.4) | 0.98 (13.4) | 1.01 (14.3) | 1.00 (13.9)

14. Secondary Outcome: Change in Triglycerides - Ratio to Baseline
Description: Change from baseline (week 0) in triglycerides (mmol/L) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Ratio of triglycerides
  Week 26: number analyzed (Participants) | 176 | 172 | 170 | 175
  Week 26 | 0.97 (41.5) | 0.92 (33.0) | 0.91 (44.8) | 0.99 (34.9)
  Week 52: number analyzed (Participants) | 172 | 167 | 167 | 169
  Week 52 | 0.93 (48.7) | 0.94 (34.9) | 0.86 (43.7) | 0.97 (39.2)

15. Secondary Outcome: Change in Total Daily Insulin Dose
Description: Change from baseline in total daily insulin dose to week 26 and week 52 is presented. Results are based on the data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units/day
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Units/day
  Week 26: number analyzed (Participants) | 178 | 173 | 173 | 178
  Week 26 | -5 (22) | -9 (21) | -8 (19) | -2 (15)
  Week 52: number analyzed (Participants) | 174 | 172 | 172 | 174
  Week 52 | 1 (26) | -8 (64) | -5 (19) | 8 (24)

16. Secondary Outcome: Participants Who Achieve: HbA1c < 7.0% (53 mmol/Mol) (American Diabetes Association (ADA) Target) (Yes/no)
Description: Number of particpants achieving HbA1c < 7.0 % (53 mmol/mol) according to American Diabetes Association (ADA) target, at week 26 and week 52. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Participants
  Week 26: number analyzed (Participants) | 176 | 174 | 173 | 176
  Week 26: Yes | 50 | 74 | 101 | 12
  Week 26: No | 126 | 100 | 72 | 164
  Week 52: number analyzed (Participants) | 173 | 169 | 168 | 172
  Week 52: Yes | 50 | 67 | 91 | 16
  Week 52: No | 123 | 102 | 77 | 156

17. Secondary Outcome: Participants Who Achieve: HbA1c ≤ 6.5% (48 mmol/Mol) (AACE Target) (Yes/no)
Description: Number of participants achieving HbA1c ≤ 6.5% (48 mmol/mol) according to American Association of Clinical Endocrinologists (AACE) target, at week 26 and week 52. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Participants
  Week 26: number analyzed (Participants) | 176 | 174 | 173 | 176
  Week 26: Yes | 24 | 45 | 74 | 6
  Week 26: No | 152 | 129 | 99 | 170
  Week 52: number analyzed (Participants) | 173 | 169 | 168 | 172
  Week 52: Yes | 20 | 33 | 65 | 4
  Week 52: No | 153 | 136 | 103 | 168

18. Secondary Outcome: Participants Who Achieve Body Weight Loss ≥5% (Yes/no)
Description: Participants who achieved weight loss more than or equal to 5% of their baseline body weight (yes/no) at weeks 26 and 52 are presented. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Participants
  Week 26: number analyzed (Participants) | 177 | 174 | 173 | 177
  Week 26: Yes | 23 | 53 | 67 | 5
  Week 26: No | 154 | 121 | 106 | 172
  Week 52: number analyzed (Participants) | 174 | 171 | 170 | 173
  Week 52: Yes | 30 | 48 | 67 | 9
  Week 52: No | 144 | 123 | 103 | 164

19. Secondary Outcome: Participants Who Achieve Body Weight Loss ≥10% (Yes/no)
Description: Participants who achieved weight loss more than or equal to 10% of their baseline body weight (yes/no) at weeks 26 and 52 are presented. The endpoint was evaluated based on data from the in-trial observation period. In trial observation period started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any. Results are based on the data from the in-trial observation period, which started at the date of randomisation and included the period after initiatiion of of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Participants
  Week 26: number analyzed (Participants) | 177 | 174 | 173 | 177
  Week 26: Yes | 2 | 12 | 19 | 1
  Week 26: No | 175 | 162 | 154 | 176
  Week 52: number analyzed (Participants) | 174 | 171 | 170 | 173
  Week 52: Yes | 4 | 17 | 21 | 1
  Week 52: No | 170 | 154 | 149 | 172

20. Secondary Outcome: Participants Who Achieve HbA1c <7.0 % (53 mmol/Mol) Without Hypoglycaemia (Severe or BG Confirmed Symptomatic Hypoglycaemia) and no Weight Gain (Yes/no)
Description: Participants who achieved HbA1c less than 7.0 % without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain (yes/no) at weeks 26 and 52 are presented. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Participants
  Week 26: number analyzed (Participants) | 176 | 174 | 173 | 176
  Week 26: Yes | 32 | 47 | 76 | 4
  Week 26: No | 144 | 127 | 97 | 172
  Week 52: number analyzed (Participants) | 173 | 169 | 168 | 172
  Week 52: Yes | 27 | 43 | 61 | 8
  Week 52: No | 146 | 126 | 107 | 164

21. Secondary Outcome: Participants Who Achieve HbA1c Reduction ≥1% (10.9 mmol/Mol) and Weight Loss ≥3% (Yes/no)
Description: Participants who achieved HbA1c reduction more than or equal to 1% of their baseline HbA1c and weight loss of more than or equal to 3% of their baseline body weight (yes/no) at weeks 26 and 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26, week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Participants
  Week 26: number analyzed (Participants) | 176 | 174 | 173 | 176
  Week 26: Yes | 28 | 51 | 76 | 7
  Week 26: No | 148 | 123 | 97 | 169
  Week 52: number analyzed (Participants) | 173 | 169 | 168 | 172
  Week 52: Yes | 20 | 37 | 64 | 5
  Week 52: No | 153 | 132 | 104 | 167

22. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the periods, from week 0 to week 26 and week 0 to week 52. Additional anti-diabetic medication was defined as use of new anti-diabetic medication for more than 21 days with the initiation at or after randomisation (week 0) and before (planned) end-of-treatment (week 52), and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Participants
  Week 0-26 | 9 | 8 | 8 | 11
  Week 0-52 | 61 | 45 | 44 | 75
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment, strata, interaction strata, and region as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0627, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.53 to 1.02]
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment, strata, and region as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0083, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.44 to 0.89]
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 22, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0019, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.40 to 0.81]

23. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime during the periods, from week 0 to week 26 and week 0 to week 52. Rescue medication was defined as use of new anti-diabetic medication as add-on to trial product and used for more than 21 days with the initiation at or after randomisation (week 1) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Participants
  Week 0-26 | 5 | 2 | 4 | 9
  Week 0-52 | 54 | 33 | 31 | 67
Statistical Analysis 1: Comparison: Oral Semaglutide 3 mg vs Placebo; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment, strata, interaction strata, and region as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.1210, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.53 to 1.08]
Statistical Analysis 2: Comparison: Oral Semaglutide 7 mg vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0007, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.32 to 0.74]
Statistical Analysis 3: Comparison: Oral Semaglutide 14 mg vs Placebo; [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p = 0.0006, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.31 to 0.73]

24. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) During Exposure to Trial Product
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 57 (52-week treatment period plus the 5-week follow-up period). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Events | 626 | 555 | 586 | 464

25. Secondary Outcome: Number of Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during week 0 to week 57 (52-week treatment period plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a subject was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Weeks 0-57
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Episodes | 196 | 180 | 147 | 156

26. Secondary Outcome: Participants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes
Description: as for outcome 25
Time Frame: Weeks 0-57
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Participants | 52 | 47 | 48 | 54

27. Secondary Outcome: Change in Amylase - Ratio to Baseline
Description: Change from baseline (week 0) in amylase (units/litre (U/L)) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Ratio of amylase
  Week 26: number analyzed (Participants) | 168 | 157 | 148 | 169
  Week 26 | 1.08 (25.4) | 1.12 (24.7) | 1.14 (26.7) | 1.01 (20.6)
  Week 52: number analyzed (Participants) | 155 | 144 | 140 | 161
  Week 52 | 1.07 (24.6) | 1.11 (26.5) | 1.17 (21.6) | 0.99 (23.5)

28. Secondary Outcome: Change in Lipase - Ratio to Baseline
Description: Change from baseline (week 0) in lipase (units/litre (U/L)) at weeks 26 and 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication
Time Frame: Week 0, week 26, week 52
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Ratio of lipase
  Week 26: number analyzed (Participants) | 168 | 157 | 148 | 169
  Week 26 | 1.14 (56.7) | 1.34 (59.1) | 1.35 (65.1) | 0.99 (47.1)
  Week 52: number analyzed (Participants) | 155 | 144 | 140 | 161
  Week 52 | 1.09 (57.5) | 1.25 (59.8) | 1.35 (49.6) | 0.99 (53.3)

29. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated at weeks 26 and 52 Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Beats/minute
  Week 26: number analyzed (Participants) | 168 | 159 | 150 | 171
  Week 26 | 1 (9) | 2 (9) | 3 (10) | -0 (9)
  Week 52: number analyzed (Participants) | 156 | 148 | 142 | 162
  Week 52 | -0 (8) | 1 (9) | 2 (10) | 0 (9)

30. Secondary Outcome: Change in SBP and DBP
Description: Change from baseline (week 0) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated at weeks 26 and 52 Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
mmHg
  SBP: Week 26: number analyzed (Participants) | 168 | 159 | 150 | 171
  SBP: Week 26 | -1 (12) | -3 (17) | -5 (14) | 1 (14)
  SBP: Week 52: number analyzed (Participants) | 156 | 148 | 142 | 162
  SBP: Week 52 | -1 (12) | -3 (16) | -6 (14) | 0 (14)
  DBP: Week 26: number analyzed (Participants) | 168 | 159 | 150 | 171
  DBP: Week 26 | -0 (8) | -1 (10) | -1 (9) | 0 (8)
  DBP: Week 52: number analyzed (Participants) | 156 | 148 | 142 | 162
  DBP: Week 52 | -1 (8) | -2 (9) | -2 (9) | -0 (8)

31. Secondary Outcome: Change in ECG Evaluation
Description: Change from baseline (week 0) in electrocardiogram (ECG) was evaluated at weeks 26 and 52. Change from baseline results are presented as shift in findings (normal; abnormal and not clinically significant (NCS); abnormal and clinically significant (CS)) from week 0 to week 26 and 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Participants
  Normal (week 0) to Normal (week 26): number analyzed (Participants) | 111 | 110 | 107 | 105
  Normal (week 0) to Normal (week 26) | 101 | 98 | 90 | 93
  Normal (week 0) to Abnormal NCS (week 26): number analyzed (Participants) | 111 | 110 | 107 | 105
  Normal (week 0) to Abnormal NCS (week 26) | 10 | 12 | 17 | 12
  Normal (week 0) to Abnormal CS (week 26): number analyzed (Participants) | 111 | 110 | 107 | 105
  Normal (week 0) to Abnormal CS (week 26) | 0 | 0 | 0 | 0
  Abnormal NCS (week 0) to Normal (week 26): number analyzed (Participants) | 66 | 59 | 63 | 70
  Abnormal NCS (week 0) to Normal (week 26) | 22 | 17 | 16 | 19
  Abnormal NCS (week 0) to Abnormal NCS (week 26): number analyzed (Participants) | 66 | 59 | 63 | 70
  Abnormal NCS (week 0) to Abnormal NCS (week 26) | 44 | 42 | 47 | 51
  Abnormal NCS (week 0) to Abnormal CS (week 26): number analyzed (Participants) | 66 | 59 | 63 | 70
  Abnormal NCS (week 0) to Abnormal CS (week 26) | 0 | 0 | 0 | 0
  Abnormal CS (week 0) to Normal (week 26): number analyzed (Participants) | 0 | 4 | 3 | 2
  Abnormal CS (week 0) to Normal (week 26) | 0 | 0 | 1 | 1
  Abnormal CS (week 0) to Abnormal NCS (week 26): number analyzed (Participants) | 0 | 4 | 3 | 2
  Abnormal CS (week 0) to Abnormal NCS (week 26) | 0 | 0 | 1 | 0
  Abnormal CS (week 0) to Abnormal CS (week 26): number analyzed (Participants) | 0 | 4 | 3 | 2
  Abnormal CS (week 0) to Abnormal CS (week 26) | 0 | 4 | 1 | 1
  Normal (week 0) to Normal (week 52): number analyzed (Participants) | 111 | 108 | 106 | 102
  Normal (week 0) to Normal (week 52) | 95 | 91 | 85 | 84
  Normal (week 0) to Abnormal NCS (week 52): number analyzed (Participants) | 111 | 108 | 106 | 102
  Normal (week 0) to Abnormal NCS (week 52) | 14 | 15 | 20 | 17
  Normal (week 0) to Abnormal CS (week 52): number analyzed (Participants) | 111 | 108 | 106 | 102
  Normal (week 0) to Abnormal CS (week 52) | 2 | 2 | 1 | 1
  Abnormal NCS to Normal (Week 52): number analyzed (Participants) | 63 | 58 | 61 | 69
  Abnormal NCS to Normal (Week 52) | 13 | 17 | 19 | 21
  Abnormal NCS to Abnormal NCS (Week 52): number analyzed (Participants) | 63 | 58 | 61 | 69
  Abnormal NCS to Abnormal NCS (Week 52) | 50 | 40 | 42 | 47
  Abnormal NCS to Abnormal CS (Week 52): number analyzed (Participants) | 63 | 58 | 61 | 69
  Abnormal NCS to Abnormal CS (Week 52) | 0 | 1 | 0 | 1
  Abnormal CS to Normal (Week 52): number analyzed (Participants) | 0 | 4 | 3 | 2
  Abnormal CS to Normal (Week 52) | 0 | 0 | 0 | 0
  Abnormal CS to Abnormal NCS (Week 52): number analyzed (Participants) | 0 | 4 | 3 | 2
  Abnormal CS to Abnormal NCS (Week 52) | 0 | 0 | 2 | 1
  Abnormal CS to Abnormal CS (Week 52): number analyzed (Participants) | 0 | 4 | 3 | 2
  Abnormal CS to Abnormal CS (Week 52) | 0 | 4 | 1 | 1

32. Secondary Outcome: Change in Physical Examination
Description: Participants with physical examination findings, normal, abnormal NCS and abnormal CS at baseline (weeks -2) and weeks 52 presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. Results are presented for the following examinations: 1) Cardiovascular system; 2) Central and peripheral nervous system; 3) Gastrointestinal system, incl. mouth; 4) General appearance; 5) Head, ears, eyes, nose, throat, neck; 6) Lymph node palpation; 7) Musculoskeletal system; 8) Respiratory system; 9) Skin; 10) Thyroid gland.
Time Frame: Week -2, week 52
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Participants
  1) Cardiovascular system (week -2): Normal | 166 | 166 | 157 | 170
  1) Cardiovascular system (week -2): Abnormal NCS | 18 | 15 | 24 | 14
  1) Cardiovascular system (week -2): Abnormal CS | 0 | 0 | 0 | 0
  1) Cardiovascular system (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  1) Cardiovascular system (week 52): Normal | 157 | 158 | 145 | 160
  1) Cardiovascular system (week 52): Abnormal NCS | 17 | 12 | 24 | 12
  1) Cardiovascular system (week 52): Abnormal CS | 0 | 0 | 1 | 1
  2) Central and peripheral nervous system (week -2): Normal | 158 | 157 | 158 | 163
  2) Central and peripheral nervous system (week -2): Abnormal NCS | 26 | 24 | 21 | 21
  2) Central and peripheral nervous system (week -2): Abnormal CS | 0 | 0 | 2 | 0
  2) Central and peripheral nervous system (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  2) Central and peripheral nervous system (week 52): Normal | 149 | 150 | 147 | 155
  2) Central and peripheral nervous system (week 52): Abnormal NCS | 25 | 20 | 22 | 18
  2) Central and peripheral nervous system (week 52): Abnormal CS | 0 | 0 | 1 | 0
  3) Gastrointestinal system, incl. mouth (week -2): Normal | 173 | 175 | 177 | 180
  3) Gastrointestinal system, incl. mouth (week -2): Abnormal NCS | 11 | 6 | 4 | 4
  3) Gastrointestinal system, incl. mouth (week -2): Abnormal CS | 0 | 0 | 0 | 0
  3) Gastrointestinal system, incl. mouth (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  3) Gastrointestinal system, incl. mouth (week 52): Normal | 163 | 164 | 166 | 171
  3) Gastrointestinal system, incl. mouth (week 52): Abnormal NCS | 9 | 6 | 3 | 1
  3) Gastrointestinal system, incl. mouth (week 52): Abnormal CS | 2 | 0 | 1 | 1
  4) General appearance (week -2): Normal | 159 | 162 | 160 | 162
  4) General appearance (week -2): Abnormal NCS | 25 | 18 | 21 | 22
  4) General appearance (week -2): Abnormal CS | 0 | 1 | 0 | 0
  4) General appearance (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  4) General appearance (week 52): Normal | 151 | 148 | 153 | 152
  4) General appearance (week 52): Abnormal NCS | 23 | 21 | 17 | 21
  4) General appearance (week 52): Abnormal CS | 0 | 1 | 0 | 0
  5) Head, ears, eyes, nose, throat, neck (week -2): Normal | 168 | 173 | 172 | 178
  5) Head, ears, eyes, nose, throat, neck (week -2): Abnormal NCS | 15 | 8 | 7 | 5
  5) Head, ears, eyes, nose, throat, neck (week -2): Abnormal CS | 1 | 0 | 2 | 1
  5) Head, ears, eyes, nose, throat, neck (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  5) Head, ears, eyes, nose, throat, neck (week 52): Normal | 161 | 164 | 165 | 166
  5) Head, ears, eyes, nose, throat, neck (week 52): Abnormal NCS | 13 | 6 | 3 | 5
  5) Head, ears, eyes, nose, throat, neck (week 52): Abnormal CS | 0 | 0 | 2 | 2
  6) Lymph node palpation (week -2): Normal | 184 | 181 | 181 | 184
  6) Lymph node palpation (week -2): Abnormal NCS | 0 | 0 | 0 | 0
  6) Lymph node palpation (week -2): Abnormal CS | 0 | 0 | 0 | 0
  6) Lymph node palpation (week 52): number analyzed (Participants) | 172 | 170 | 170 | 173
  6) Lymph node palpation (week 52): Normal | 172 | 170 | 170 | 172
  6) Lymph node palpation (week 52): Abnormal NCS | 0 | 0 | 0 | 1
  6) Lymph node palpation (week 52): Abnormal CS | 0 | 0 | 0 | 0
  7) Musculoskeletal system (week -2): Normal | 171 | 170 | 169 | 175
  7) Musculoskeletal system (week -2): Abnormal NCS | 13 | 10 | 9 | 9
  7) Musculoskeletal system (week -2): Abnormal CS | 0 | 1 | 3 | 0
  7) Musculoskeletal system (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  7) Musculoskeletal system (week 52): Normal | 160 | 160 | 159 | 164
  7) Musculoskeletal system (week 52): Abnormal NCS | 11 | 9 | 8 | 8
  7) Musculoskeletal system (week 52): Abnormal CS | 3 | 1 | 3 | 1
  8) Respiratory system (week -2): Normal | 182 | 177 | 180 | 184
  8) Respiratory system (week -2): Abnormal NCS | 1 | 4 | 1 | 0
  8) Respiratory system (week -2): Abnormal CS | 1 | 0 | 0 | 0
  8) Respiratory system (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  8) Respiratory system (week 52): Normal | 173 | 164 | 170 | 173
  8) Respiratory system (week 52): Abnormal NCS | 1 | 6 | 0 | 0
  8) Respiratory system (week 52): Abnormal CS | 0 | 0 | 0 | 0
  9) Skin (week -2): Normal | 156 | 153 | 159 | 162
  9) Skin (week -2): Abnormal NCS | 27 | 28 | 22 | 21
  9) Skin (week -2): Abnormal CS | 1 | 0 | 0 | 1
  9) Skin (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  9) Skin (week 52): Normal | 152 | 144 | 151 | 155
  9) Skin (week 52): Abnormal NCS | 20 | 26 | 18 | 18
  9) Skin (week 52): Abnormal CS | 2 | 0 | 1 | 0
  10) Thyroid gland (week -2): Normal | 177 | 176 | 176 | 177
  10) Thyroid gland (week -2): Abnormal NCS | 7 | 5 | 5 | 5
  10) Thyroid gland (week -2): Abnormal CS | 0 | 0 | 0 | 2
  10) Thyroid gland (week 52): number analyzed (Participants) | 174 | 170 | 170 | 173
  10) Thyroid gland (week 52): Normal | 166 | 165 | 168 | 166
  10) Thyroid gland (week 52): Abnormal NCS | 8 | 5 | 2 | 6
  10) Thyroid gland (week 52): Abnormal CS | 0 | 0 | 0 | 1

33. Secondary Outcome: Change in Eye Examination Category
Description: Participants with eye examination (fundoscopy) findings, normal, abnormal NCS and abnormal CS at baseline (week -2) and week 52 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week -2, week 52
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 181 | 181 | 184
Participants
  Left eye (week -2): number analyzed (Participants) | 184 | 180 | 181 | 184
  Left eye (week -2): Normal | 89 | 102 | 99 | 108
  Left eye (week -2): Abnormal NCS | 76 | 64 | 64 | 55
  Left eye (week -2): Abnormal CS | 19 | 14 | 18 | 21
  Left eye (week 52): number analyzed (Participants) | 170 | 167 | 162 | 166
  Left eye (week 52): Normal | 83 | 102 | 92 | 88
  Left eye (week 52): Abnormal NCS | 65 | 51 | 52 | 53
  Left eye (week 52): Abnormal CS | 22 | 14 | 18 | 25
  Right eye (week -2): number analyzed (Participants) | 184 | 180 | 181 | 184
  Right eye (week -2): Normal | 85 | 104 | 99 | 106
  Right eye (week -2): Abnormal NCS | 76 | 63 | 64 | 58
  Right eye (week -2): Abnormal CS | 23 | 13 | 18 | 20
  Right eye (week 52): number analyzed (Participants) | 169 | 167 | 163 | 166
  Right eye (week 52): Normal | 79 | 99 | 97 | 90
  Right eye (week 52): Abnormal NCS | 67 | 54 | 51 | 50
  Right eye (week 52): Abnormal CS | 23 | 14 | 15 | 26

34. Secondary Outcome: Semaglutide Plasma Concentrations for Population PK Analyses
Description: This outcome measure is only applicable for the oral semaglutide treatment arms (3 mg, 7 mg and 14 mg). Semaglutide plasma concentrations were measured at week 4, 14, 26, 38 and 52. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-52
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg
Number analyzed (Participants) | 184 | 182 | 181
nmol/L
  Week 4: number analyzed (Participants) | 177 | 176 | 170
  Week 4 | 2.9 (111.2) | 2.9 (116.4) | 2.9 (98.1)
  Week 14: number analyzed (Participants) | 172 | 161 | 155
  Week 14 | 2.9 (106.9) | 7.5 (143.2) | 14.5 (172.7)
  Week 26: number analyzed (Participants) | 167 | 160 | 148
  Week 26 | 2.7 (124.7) | 7.2 (141.4) | 12.6 (203.9)
  Week 38: number analyzed (Participants) | 161 | 150 | 143
  Week 38 | 2.5 (123.8) | 6.9 (139.7) | 10.8 (238.3)
  Week 52: number analyzed (Participants) | 154 | 148 | 142
  Week 52 | 2.4 (126.0) | 5.8 (160.5) | 11.9 (210.4)

35. Secondary Outcome: Change in SF-36v2 (Acute Version) Health Survey: Scores From the 8 Domains, the Physical Component Summary (PCS) and the Mental Component Summary (MCS)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at weeks 26 and 52. A positive change score indicates an improvement since baseline. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Score on a scale
  1) Physical functioning (Week 26): number analyzed (Participants) | 178 | 172 | 173 | 176
  1) Physical functioning (Week 26) | 0.53 (7.58) | 0.52 (6.61) | -0.07 (6.75) | -0.82 (7.25)
  1) Physical functioning (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  1) Physical functioning (Week 52) | 0.51 (8.27) | -0.40 (6.69) | -0.32 (7.55) | -0.77 (6.31)
  2) Role Physical (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  2) Role Physical (Week 26) | -0.32 (8.64) | -0.43 (8.45) | 0.04 (6.81) | -0.39 (7.19)
  2) Role Physical (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  2) Role Physical (Week 52) | 0.00 (8.46) | -0.76 (7.88) | -0.87 (7.97) | -0.93 (8.28)
  3) Bodily Pain (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  3) Bodily Pain (Week 26) | -0.02 (9.75) | 1.47 (8.98) | -0.18 (7.76) | -0.72 (9.88)
  3) Bodily Pain (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  3) Bodily Pain (Week 52) | -0.40 (9.78) | 0.56 (9.70) | -0.21 (8.22) | -0.64 (11.23)
  4) General Health (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  4) General Health (Week 26) | 1.43 (6.75) | 0.70 (7.23) | 1.26 (6.11) | -0.36 (6.35)
  4) General Health (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  4) General Health (Week 52) | 0.92 (6.27) | 0.75 (7.00) | 1.38 (6.04) | -1.43 (6.95)
  5) Vitality (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  5) Vitality (Week 26) | -0.56 (7.73) | -1.27 (6.70) | 0.14 (8.01) | -1.69 (7.18)
  5) Vitality (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  5) Vitality (Week 52) | -0.53 (8.24) | -1.43 (7.68) | 0.70 (8.40) | -1.09 (7.12)
  6) Social functioning (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  6) Social functioning (Week 26) | -0.31 (8.86) | 0.34 (8.65) | -0.51 (9.25) | -1.10 (8.03)
  6) Social functioning (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  6) Social functioning (Week 52) | 0.11 (9.73) | -0.61 (10.09) | 0.03 (8.73) | -1.74 (8.70)
  7) Role emotional (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  7) Role emotional (Week 26) | -0.94 (11.20) | 0.62 (9.94) | 0.24 (9.78) | -1.50 (9.08)
  7) Role emotional (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  7) Role emotional (Week 52) | 0.77 (10.61) | -0.34 (10.58) | 0.09 (9.91) | -2.78 (10.81)
  8) Mental health (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  8) Mental health (Week 26) | -1.41 (9.29) | -0.82 (7.58) | 0.99 (8.50) | -2.32 (7.57)
  8) Mental health (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  8) Mental health (Week 52) | -0.48 (8.69) | -0.74 (9.91) | 0.89 (8.39) | -1.30 (8.00)
  9) Physical component summary (Week 26): number analyzed (Participants) | 178 | 172 | 173 | 176
  9) Physical component summary (Week 26) | 0.94 (6.20) | 0.75 (6.27) | -0.02 (4.81) | -0.05 (6.07)
  9) Physical component summary (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  9) Physical component summary (Week 52) | 0.26 (6.78) | 0.12 (6.24) | -0.36 (6.09) | -0.41 (6.54)
  10) Mental component summary (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  10) Mental component summary (Week 26) | -1.41 (9.50) | -0.55 (7.91) | 0.49 (8.72) | -2.16 (7.45)
  10) Mental component summary (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  10) Mental component summary (Week 52) | -0.09 (8.45) | -0.89 (9.66) | 0.82 (8.57) | -2.19 (8.23)

36. Secondary Outcome: Change in IWQoL-Lite-CT: Total Score and Scores From the 4 Domains
Description: The Impact of Weight on Quality of Life Clinical Trials Version (IWQOL-Lite-CT) is designed to assess the impact of changes in weight on patients' quality of life within the context of clinical trials. The items of the IWQOL-Lite-CT pertain to physical functioning (physical, physical function and pain/discomfort) and psychosocial domains and all items employ a 5-point graded response scale (never, rarely, sometimes, usually, always; or not at all true, a little true, moderately true, mostly true, completely true). All IWQOL-Lite-CT composite scores range from 0 to 100, with higher scores reflecting better levels of functioning. Results are based on the data from the in-trial observation period, which started at the date of randomisation and included the period after initiation of rescue medication and/or premature trial product discontinuation, if any.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Score on a scale
  1) Psychosocial (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  1) Psychosocial (Week 26) | 1.45 (13.89) | -0.32 (13.58) | 4.10 (14.24) | -0.49 (11.62)
  1) Psychosocial (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  1) Psychosocial (Week 52) | 1.96 (14.89) | -0.92 (13.20) | 5.35 (15.89) | -0.46 (14.46)
  2) Physical (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  2) Physical (Week 26) | 2.29 (17.30) | -0.66 (15.20) | 2.15 (14.66) | -1.75 (13.28)
  2) Physical (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  2) Physical (Week 52) | 3.10 (18.81) | -0.53 (15.30) | 2.50 (15.33) | -1.24 (16.36)
  3) Physical function(Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  3) Physical function(Week 26) | 1.88 (18.64) | -0.35 (16.28) | 2.51 (15.94) | -1.70 (15.12)
  3) Physical function(Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  3) Physical function(Week 52) | 3.45 (19.79) | -0.59 (15.85) | 2.59 (16.02) | -0.98 (17.33)
  4) Pain/discomfort (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  4) Pain/discomfort (Week 26) | 3.30 (22.52) | -1.45 (21.22) | 1.23 (22.86) | -1.85 (21.51)
  4) Pain/discomfort (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  4) Pain/discomfort (Week 52) | 2.23 (24.48) | -0.37 (20.88) | 2.28 (22.12) | -1.88 (22.48)
  5) IWQOL-Lite-CT Total (Week 26): number analyzed (Participants) | 178 | 173 | 173 | 176
  5) IWQOL-Lite-CT Total (Week 26) | 1.74 (13.37) | -0.45 (12.47) | 3.41 (12.19) | -0.94 (10.40)
  5) IWQOL-Lite-CT Total (Week 52): number analyzed (Participants) | 174 | 169 | 170 | 173
  5) IWQOL-Lite-CT Total (Week 52) | 2.35 (14.50) | -0.79 (12.47) | 4.35 (13.82) | -0.73 (13.50)

37. Secondary Outcome: Change in DTSQs: Individual Items and Treatment Satisfaction Score (6 of the 8 Items Summed)
Description: Change from baseline (week 0) in Diabetes Treatment Satisfaction Questionnaire - status version (DTSQs) was evaluated at week 26 and week 52. The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items 1, 4 -8. For items 2 and 3 a higher score indicates a higher patient perceived experience of hyperglycaemia and hypoglycaemia, respectively. Thus, lower scores indicate a perception of blood glucose levels being "none of the time" unacceptably high (item 2) or low (item 3). The domain score of total treatment satisfaction (total treatment satisfaction score) was computed by adding the six items scores 1, 4-8. The score has a minimum of 0 and a maximum of 36. A higher treatment satisfaction score indicates a higher level of treatment satisfaction.
Time Frame: Week 0, week 26, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 184 | 182 | 181 | 184
Score on a scale
  Satisfaction with treatment: wk 26: number analyzed (Participants) | 178 | 172 | 173 | 176
  Satisfaction with treatment: wk 26 | 0.47 (1.27) | 0.59 (1.49) | 0.63 (1.50) | 0.18 (1.40)
  Satisfaction with treatment: wk 52: number analyzed (Participants) | 174 | 169 | 169 | 173
  Satisfaction with treatment: wk 52 | 0.53 (1.42) | 0.51 (1.45) | 0.78 (1.53) | 0.20 (1.17)
  Feeling of unacceptably high blood sugars: wk 26: number analyzed (Participants) | 178 | 172 | 173 | 176
  Feeling of unacceptably high blood sugars: wk 26 | -0.62 (1.89) | -1.23 (1.98) | -1.29 (1.96) | -0.28 (1.85)
  Feeling of unacceptably high blood sugars: wk 52: number analyzed (Participants) | 174 | 169 | 170 | 173
  Feeling of unacceptably high blood sugars: wk 52 | -0.70 (2.02) | -1.15 (1.95) | -1.34 (2.13) | -0.41 (1.91)
  Feeling of unacceptably low blood sugars: wk 26: number analyzed (Participants) | 177 | 172 | 173 | 176
  Feeling of unacceptably low blood sugars: wk 26 | 0.07 (1.97) | -0.06 (1.70) | 0.13 (2.08) | -0.15 (1.91)
  Feeling of unacceptably low blood sugars: wk 52: number analyzed (Participants) | 174 | 168 | 170 | 173
  Feeling of unacceptably low blood sugars: wk 52 | 0.04 (1.90) | -0.10 (1.74) | -0.06 (2.04) | -0.02 (1.80)
  Convenience of treatment: wk 26: number analyzed (Participants) | 178 | 172 | 173 | 176
  Convenience of treatment: wk 26 | 0.51 (1.25) | 0.50 (1.68) | 0.50 (1.43) | 0.20 (1.49)
  Convenience of treatment: wk 52: number analyzed (Participants) | 174 | 169 | 169 | 173
  Convenience of treatment: wk 52 | 0.38 (1.50) | 0.52 (1.54) | 0.44 (1.70) | 0.19 (1.50)
  Flexibility of treatment: wk 26: number analyzed (Participants) | 178 | 172 | 173 | 176
  Flexibility of treatment: wk 26 | 0.31 (1.43) | 0.37 (1.66) | 0.40 (1.43) | 0.23 (1.34)
  Flexibility of treatment: wk 52: number analyzed (Participants) | 174 | 169 | 169 | 173
  Flexibility of treatment: wk 52 | 0.25 (1.60) | 0.42 (1.58) | 0.46 (1.53) | 0.23 (1.54)
  Satisfaction with understading of diabetes: wk 26: number analyzed (Participants) | 178 | 172 | 173 | 176
  Satisfaction with understading of diabetes: wk 26 | 0.24 (1.31) | 0.31 (1.40) | 0.27 (1.22) | 0.04 (0.94)
  Satisfaction with understading of diabetes: wk 52: number analyzed (Participants) | 174 | 169 | 170 | 173
  Satisfaction with understading of diabetes: wk 52 | 0.25 (1.40) | 0.35 (1.45) | 0.34 (1.28) | 0.03 (1.18)
  Recommending treatment to others: wk 26: number analyzed (Participants) | 178 | 172 | 173 | 176
  Recommending treatment to others: wk 26 | 0.20 (1.50) | 0.66 (1.79) | 0.53 (1.53) | 0.02 (1.40)
  Recommending treatment to others: wk 52: number analyzed (Participants) | 174 | 169 | 170 | 173
  Recommending treatment to others: wk 52 | 0.32 (1.47) | 0.63 (1.55) | 0.65 (1.62) | -0.01 (1.34)
  Satisfaction to continue present treatment: wk 26: number analyzed (Participants) | 177 | 172 | 173 | 176
  Satisfaction to continue present treatment: wk 26 | 0.40 (1.30) | 0.57 (1.65) | 0.58 (1.39) | 0.09 (1.24)
  Satisfaction to continue present treatment: wk 52: number analyzed (Participants) | 174 | 169 | 169 | 172
  Satisfaction to continue present treatment: wk 52 | 0.41 (1.27) | 0.56 (1.58) | 0.65 (1.52) | 0.03 (1.35)
  Total treatment satisfaction: wk 26: number analyzed (Participants) | 178 | 172 | 173 | 176
  Total treatment satisfaction: wk 26 | 2.12 (5.38) | 3.00 (7.36) | 2.90 (5.95) | 0.76 (5.52)
  Total treatmemt satisfaction: wk 52: number analyzed (Participants) | 174 | 169 | 169 | 173
  Total treatmemt satisfaction: wk 52 | 2.14 (6.02) | 2.99 (6.80) | 3.32 (6.78) | 0.67 (5.92)

ADVERSE EVENTS:
Time Frame: Week 0 to week 57 (52 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 3 mg: Subjects were to take oral semaglutide 3 mg tablets once daily from week 1 to 52.
- Oral Semaglutide 7 mg: Subjects were to take oral semaglutide tablets once daily in a dose escalation manner from week 1 to 52: 3 mg from week 1 to 4 and 7 mg from week 5 to 52.
- Oral Semaglutide 14 mg: Subjects were to take oral semaglutide tablets once daily in a dose escalation manner from week 1 to 52: 3 mg from week 1 to 4, 7 mg from week 5 to 8 and 14 mg from week 9 to 52.
Arm/Group | Oral Semaglutide 3 mg | Oral Semaglutide 7 mg | Oral Semaglutide 14 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/181 | 3/181 | 0/184
Serious Adverse Events (participants affected / at risk) | 25/184 | 19/181 | 12/181 | 17/184
Other Adverse Events (participants affected / at risk) | 77/184 | 86/181 | 100/181 | 73/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=184) | Oral Semaglutide 7 mg (N=181) | Oral Semaglutide 14 mg (N=181) | Placebo (N=184)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mononeuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal myelogram (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White matter lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 3 mg (N=184) | Oral Semaglutide 7 mg (N=181) | Oral Semaglutide 14 mg (N=181) | Placebo (N=184)
Abdominal discomfort (Gastrointestinal disorders) | 7 (8) | 11 (12) | 10 (11) | 3 (3)
Constipation (Gastrointestinal disorders) | 8 (8) | 15 (16) | 12 (13) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 18 (19) | 23 (24) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 16 (19) | 22 (26) | 26 (40) | 11 (15)
Hypertension (Vascular disorders) | 3 (4) | 4 (4) | 1 (1) | 11 (12)
Nasopharyngitis (Infections and infestations) | 27 (42) | 21 (32) | 18 (29) | 27 (35)
Nausea (Gastrointestinal disorders) | 21 (23) | 30 (34) | 41 (60) | 13 (19)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 6 (8) | 13 (13) | 13 (17)
Urinary tract infection (Infections and infestations) | 6 (10) | 5 (6) | 10 (10) | 7 (12)
Vomiting (Gastrointestinal disorders) | 11 (14) | 14 (17) | 17 (28) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT03021187/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT03021187/SAP_001.pdf